CLINICAL TRIAL: NCT02860065
Title: Phase II, Modified Single-Blind, Sequential Treatment, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Cerebral Efficacy of CPC-201 in Patients With Alzheimer's Disease Type Dementia: PET Study
Brief Title: CPC-201 Alzheimer's Disease Type Dementia: PET Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Chase Pharmaceuticals Corporation, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPC-001-15
Record Dates: First submitted 2016-07-26; First posted 2016-08-09 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPC-201 (Experimental): combination of solifenacin and high doses of donepezil
  Interventions: Drug: CPC-201; Other: Positron emission tomography (PET)

INTERVENTIONS:
Drug: CPC-201 — solifenacin and donepezil
Other: Positron emission tomography (PET) — measure activity of cerebral acetylcholinesterase

SUMMARY:
The purpose of this study is to compare the effect of low and high dose CPC-201 on brain function including cerebral acetylcholinesterase (AChE) activity measured by positron emission tomography (PET).

DETAILED DESCRIPTION:
Patients will continue on the 10 mg/day dose of donepezil with the addition of 15 mg/day of solifenacin at least for a week, donepezil will be titrated from 10 to 50 mg/day (maximum allowed dose; MAD) or each patient's MTD with increments of 5 or 10 mg weekly or bi-weekly as medically appropriate. When the MTD or MAD of donepezil co-administered with solifenacin 15 mg/day as CPC-201 has been reached, treatment will be stably maintained, as tolerated, for 3 months.

Patients successfully completing this protocol will have the option of continuing in an open extension of their CPC-201 treatment (separate protocol) or returned to their pre-admission therapeutic regimen and discharged from the study.

On the days of study drug dose increase, patients will be evaluated at a clinic as an out-patient.

This is a sequential study conducted in 6 phases in AD patients who had previously been receiving donepezil at a dose of 10 mg/day:

1. Screening
2. Baseline assessment
3. Solifenacin introduction at a dose of 15 mg/day (given with continued donepezil 10 mg/day as CPC-201);
4. Donepezil dose escalation to each subject's MTD or 50 mg/day (MAD), given in combination with solifenacin 15 mg/day as CPC-201;
5. Donepezil maintenance at its MTD (or MAD) combined with solifenacin 15 mg/day as CPC-201 for 3 months;
6. Protocol exit (after resumption of pre-study treatment regimen and successful completion of a one month post-study safety check) or optional entry into a 6 month extension phase.

Baseline assessment (during solifenacin introduction): Upon successful completion of a screening evaluation and entry into this study, participants will continue to receive 10 mg donepezil and receive neuropsychological evaluations at the clinic together with a 11C-PMP PET scan and associated MRI studies of the brain in accordance with the University of Michigan.

Solifenacin introduction: After the one week baseline assessment period, solifenacin treatment will be initiated at 15 mg/day for at least one week while patients continue to receive donepezil at a dose of 10 mg/day. Those who do not tolerate solifenacin will be withdrawn from the study and replaced.

Donepezil escalation: During this phase, while continuing to receive 15 mg/day of solifenacin, the dose of donepezil will be gradually increased at weekly or bi-weekly with increments of 5 or 10 mg as tolerated. The dose of donepezil will be increased until the first intolerable dose (FID) is reached or a dose of 50 mg/day is attained, whichever comes first. Once patients reach their FID, their MTD will be defined as their immediately preceding, tolerated dose. During dose titration, investigators may extend the same donepezil dose for additional days or temporarily (or permanently) reduce it as medically indicated. On the days of donepezil dose increase, patients will remain in the clinic for at least 5 hours after study drug administration or until signs and symptoms of medically significant adverse effects abate.

Donepezil dose maintenance: During this phase, patients will continue treatment with donepezil (at MTD) and solifenacin (15 mg/day) for 3 months (± 2 weeks). All will be followed by weekly telephone interviews and monthly clinic visits to assess safety and tolerability. If intolerable adverse events (AEs) develop, the daily dose of donepezil will be down-titrated, and the patient will continue treatment on their new MTD for an additional 2 weeks or up to completion of the maintenance phase, whichever comes last. Patients who continue to experience intolerable AEs after several down-titrations will be withdrawn from the study.

End of study testing at the end of donepezil dose maintenance: After completion of 3-months (± 2 weeks) treatment with donepezil (at MTD) and solifenacin (15 mg/day), study participants will receive a repeat of their clinical examination, routine laboratory safety tests and PET associated studies.

Patients successfully completing this protocol will then have the option of continuing in an open extension of their CPC-201 treatment (separate protocol) or to be returned to their pre-admission therapeutic regimen and discharged from the study.

Study Exit: Upon termination of this study, subjects will return to their original daily donepezil dose. Investigator will decide whether the patient should discontinue high dose of donepezil without down-titration, or whether donepezil should be down-titrated to their prestudy donepezil dose. Whatever the decision, the patient will ordinarily be treated at least an additional 7 days with solifenacin 15 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an Institutional Review Board (IRB) approved informed consent document indicating that they understand the purpose of and procedures required by the study protocol and are willing to participate in the study and comply with all its procedures and restrictions. Informed consent must be obtained from the patient and/or a designated representative prior to initiating screening procedures to evaluate their eligibility for the study.
2. Aged 50 - 79 years inclusive.
3. Meet the diagnosis of probable AD consistent with:

   * Revised National Institute on Aging-Alzheimer's Association (NIA-ADA) criteria and
   * Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria.
4. Of mild to moderate severity: Mini-Mental Status Exam (MMSE) score 10 - 24 inclusive.
5. Rosen-Modified Hachinski Ischemia Score of ≤4.
6. Have a suitable caregiver to supervise the at-home administration of study drugs and observe for AEs.
7. Treated with donepezil 10 mg/day (given once daily) for at least 4 weeks just prior to study entry and to have safely tolerated, as judged clinically by the investigator.
8. Patients must be in generally good health as indicated by their medical history and physical examination, vital signs, electrocardiogram (ECG), and standard laboratory tests.

Exclusion Criteria:

1. Women of child bearing potential.
2. History or presence of a seizure disorder.
3. History of uncontrolled peptic ulcer disease, urinary or gastric retention; asthma or obstructive pulmonary disease.
4. History or presence of uncontrolled bladder outflow obstruction, gastrointestinal obstructive disorder or reduced gastrointestinal motility, or narrow-angle glaucoma.
5. Renal and hepatic dysfunction with:

   * Total Bilirubin: >1.5 x UNL
   * AST: >2.5 x UNL
   * ALT: >2.5 x UNL
   * Serum Creatinine: >1.5 x UNL
   * Creatinine Clearance: <30 mL/min (calculated by Cockcroft and Gault equation)
6. History or presence of myasthenia.
7. History of Prolonged QT Syndrome.
8. History of unexplained syncope.
9. Myocardial infarction or hospitalization for congestive heart failure within 6 months.
10. Patients has implanted cardiac pacemaker, implantable cardiac defibrillator (ICD), or metallic objects located in the eye, neck, ear, brain or blood vessel walls.
11. ECG findings of:

    * Complete Left Bundle Branch block;
    * Ventricular pacing;
    * 2nd degree or 3rd degree AV block;
    * Atrial fibrillation or atrial flutter;
    * Heart rate <45 or >100;
    * PR >220 msec; or
    * QTcF >450 msec in male, >470 msec in female
12. Patients treated with the following medications within 8 weeks of screening

    * AChEIs (other than donepezil),
    * Peripherally acting anticholinergics (such as drugs for the treatment of overactive bladder disorder),
    * Psychoactive medications (including antipsychotics, antidepressants, anxiolytics or sedative hypnotics) having significant anticholinergic effects and/or believed to affect cognitive function.

    Other medications are acceptable, at the investigators discretion, if dosage is held stable for at least 4 weeks prior to screening and throughout the study.
13. Claustrophobia
14. Patients considered unlikely to cooperate in the study, and/or poor compliance anticipated by the investigator.
15. Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives.
16. Patients who have participated in another clinical trial with an investigational drug within previous 30 days.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-30 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Donepezil Maximum tolerated dose (MTD) change on imaging | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System--West Bloomfield Hospital, West Bloomfield, Michigan, United States